CLINICAL TRIAL: NCT03878563
Title: Alterations in Intestinal Mucosal Barrier Visualized by Confocal Laser Endomicroscopy in Liver Cirrhosis: a Pilot Trial
Brief Title: Alterations in Intestinal Mucosal Barrier Visualized by Confocal Laser Endomicroscopy in Liver Cirrhosis: a Pilot Trial (AMBIC)
Acronym: AMBIC
Status: Terminated | Type: Observational
Why Stopped: Sponsor-PI left Switzerland
Sponsor: Dr.med. Monica Rusticeanu (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other); University of Bern (Other)
Responsible Party: Sponsor-Investigator, Dr.med. Monica Rusticeanu, Dr.med. M. Rusticeanu LÄ stv. Gastroenterologie und Hepatologie, Spital Limmattal Schlieren
Organization: Spital Limmattal Schlieren (Other)
Other Study IDs: 2017-00249
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Liver Cirrhoses
Keywords: intestinal barrier dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- ascites with/without SBP: Cirrhosis with ascites and existing SBP or prior SBP
  Interventions: Device: Cellvisio 100 Series (fibered confocal microscopic system)
- ascites and decreased protein concentrati: Cirrhosis with ascites and decreased protein concentration <1,5 g/d
  Interventions: Device: Cellvisio 100 Series (fibered confocal microscopic system)
- ascites and normal protein concentration: Liver cirrhosis witha scites and protein concentration >1,5 g/d
  Interventions: Device: Cellvisio 100 Series (fibered confocal microscopic system)
- Liver cirrhosis without ascites: Patients with liver corrhosis without ascites
  Interventions: Device: Cellvisio 100 Series (fibered confocal microscopic system)
- Healthy controls without liver cirrhosis or other pathology: Healthy pacients (without chronic disease) undergoing screening coloscopy or gastroscopy
  Interventions: Device: Cellvisio 100 Series (fibered confocal microscopic system)

INTERVENTIONS:
Device: Cellvisio 100 Series (fibered confocal microscopic system) — This system is intended to allow confocal laser imaging of the internal microstructure of tissues within or adjacent to anatomical tracts, i.e. Gastrointestinal accessed trough an endoscope.
  An 488-nm wavelength laser system is used, images are steamed at a frame rate of 12 frames per second, obtaining real time videos of the mucosa. In this trial we will use the Confocal miniprobe ColoFlex UHD and GastroFlex UHD.

SUMMARY:
Clinical trial with medical devices. A diagnostic trial conducted to find a better (less invasive) procedure for predicting the onset of spontaneous bacterial peritonitis(SBP), which is a complication of liver cirrhosis with ascites.The current recommendation for primary prophylaxis of SBP include a low protein content of the ascitic fluid or a gastrointestinal bleeding. This trial will use the CLE (confocal laser endomicroscopy) technic in order to quantify the intestinal permeability in patients with liver cirrhosis and correlate this to the onset of spontaneous bacterial peritonitis.We aim to evaluate a new diagnostic tool (the confocal laser endoscopy(CLE) technique -cellvizio- in the setting of endoscopy and defining parameters that are altered in cirrhotic patients of different severity and being at risk of developing a SBP (spontaneous bacterial peritonitis).The parameters assessed by confocal laser endomicroscopy will be correlated with the protein content in ascitic fluid and the patient will be monitored for time to occurrence of spontaneous bacterial peritonitis.

Defining a correlation between the quantified loss of intestinal integrity and i) total protein concentration in the ascitic fluid and ii) stadium of liver disease (Child class A, B or C)

ELIGIBILITY:
Inclusion Criteria:

Adult individual (>18yo) with liver cirrhosis of any cause and healthy controls undergoing elective endoscopy

Exclusion Criteria:

* Patients younger than < 18, older than 80 years
* Pregnant or breastfeeding women
* Known allergy to fluorescein.
* Cardiac disease
* Asthma bronchiale
* Patients with inability or unwillingness to provide blood samples or samples of ascitic fluid.
* patients unable to give informed consent
* non-resident patients
* contraindication for an endoscopic examination

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with liver cirrhosis and healthy controls, older than 18 years and younger than 80 years
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
occurrence of spontaneous bacterial peritonitis at 12 months | 24 months
  The parameters assessed by confocal laser endomicroscopy will be correlated with the protein content in ascitic fluid and the patient will be monitored for occurrence of spontaneous bacterial peritonitis for the next 12 months.

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Limmattal Spital, Schlieren, Canton of Zurich
  - Universitätsspital Bern, Bern